CLINICAL TRIAL: NCT03702504
Title: Margherita-PROSAFE:Promoting Patient Safety and Quality Improvement in Critical Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Other)
Collaborators: European Commission (Other); Friedrich Schiller University of Jena (Unknown); General Hospital of Novo mesto (Other); Intensive Care Forum (ICF) (Unknown); Medical University of Warsaw (Other); University of Nicosia (Other); Semmelweis University Budapest (Unknown); University College, London (Other); Univerzitetni Klinikni Center Ljubljana (Unknown); Ben-Gurion University of the Negev (Other); University of Crete Medical School - University Hospital of Heraklion (Unknown); Orobix Srl (Unknown)
Responsible Party: Sponsor
Other Study IDs: N° 2007331
Record Dates: First submitted 2017-12-22; First posted 2018-10-11 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Intensive Care Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general objective is to promote patient safety and quality improvement in critical care towards a significant reduction of observed mortality rates and economic costs through the improvement of outcomes and reduction of medical errors.

DETAILED DESCRIPTION:
Intensive care is one of the largest, most expensive, most complex components of European healthcare; each year about one million patients are admitted to intensive care units across Europe. The project contributes to European society in the long-term by promoting cooperation between member states in the critical care domain, with a view to improving the safety of patients admitted to ICUs and to continuously assessing performance through international comparison of outcomes and procedures. It also contributes to the exchange of good practice, reduce medical errors and promote high quality services in public health.

Patient safety and quality of care measurement and improvement are among the most important, challenging aspects of public health. The intensive and critical care domains need continuous monitoring and improvement considering the high mortality rates in and major financial investments required by ICUs. However, collection of ICU performance data is not standardized and no transnational EU project to improve patient safety and to assess performance and quality of care is currently operating for ICUs.

The project provides long-term benefits to European society by promoting cooperation between member states in the critical care domain with a view to improving the safety of patients admitted to ICUs and performing continuous performance evaluation through comparison of outcomes and procedures at international level.

The aim of this project is to export the positive results achieved through an Italian experience (Margherita system) to other European countries, addressing in particular new member states where benchmarking is sparse and uncoordinated and quality assessment and comparison is needed.

Methods and means:

It is proposed to build an ICU network across EU to collect standardized data on admitted patients, to perform statistical analyses based on national and intercountry comparisons and to appropriately identify and manage strengths and weaknesses in performance.

ELIGIBILITY:
Inclusion Criteria:

* All the patients admitted in ICU

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted in partecipating ICU
Sampling Method: Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2008-11 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | 1 year
  Hospital mortality is required to calculated different indicators:
  * SMR: it is the ratio between the mortality rate actually observed in a specific centre and the mortality that would have been expected had this centre performed according to the average of all the other participating centers, as they behaved in the same period, in the same country.
  * VLAD: it shows the performance of each individual ICU (expressed along the y axis) against time (reported on the x axis). When the plot rises, it means that in the period in question the ICU performed better than the average, in terms of lives saved, and vice versa when the plot declines, in terms of lives lost compared to the average performance.
  * GiViTI Calibration belt: it represents the confidence band that correlates the observed and the expected (according to the average performance) mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale A. Manzoni, U.O. Anestesia e Rianimazione 1, Lecco, Lombardy, Italy